CLINICAL TRIAL: NCT07396740
Title: Description of the Stroma of Solid Tumors
Brief Title: Description of the Stroma of Solid Tumors (DISTRO)
Acronym: DISTRO
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0204 - DISTRO
Record Dates: First submitted 2024-09-18; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cancer; Benign Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to describe the cellular and non-cellular components of different types of benign and malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* any patient with pathological sample analyzed in Brest UH since 2000

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: any patient with pathological sample analyzed in Brest UH since 2000
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Composition of the stroma | 5 years
  Numbers of non tumor cells per mm²
Composition of the stroma | 5 years
  Percentages of matrix within tissu areas

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement